#### STATISTICAL ANALYSIS PLAN

STUDY TITLE: Randomized, Double-Blind, Placebo-Controlled Phase 2

Study of the Efficacy and Safety of Intravenous Pamrevlumab, a Monoclonal Antibody Against Connective Tissue Growth Factor (CTGF), in

Hospitalized Patients with Acute COVID-19 Disease

PROTOCOL NUMBER: FGCL-3019-098

**Protocol Version:** Amendment 1.0

Version

**Release Date:** 4/20/2021 final

#### **CONFIDENTIALITY STATEMENT**

The information contained in this document is confidential and proprietary to FibroGen, Inc. No part of this document or any of the information contained herein may be transmitted, disclosed, shared, reproduced, published or utilized by any persons without prior written authorization by FibroGen, Inc.

# **SIGNATURE PAGE**

# **Approvals**

I have reviewed and accepted the information in this document to be a true and accurate representation of the Statistical Analysis Plan.

# **Initiator:**

| Signature: | *See appended final page for 21CFR Part 11 compliant approval | Date: |
|---|---|---|
| _ | | |
| Reviewed by: | | |
| Signature: | *See appended final page for 21CFR Part 11 compliant approval | Date: |
| _ | | |
| Signature: | *See appended final page for 21CFR Part 11 compliant approval | Date: |
| Signature: | *See appended final page for 21CFR Part 11 compliant approval | <b>Date:</b> |
| Signature: | *See appended final page for 21CFR Part 11 compliant approval | <b>Date:</b> |
| Signature: | *See appended final page for 21CFR Part 11 compliant approval | <b>Date:</b> |

# **Signature Significance**

The following significance is lent to the signatures on the Approvals page of this document.

| Signatory | Significance |
|---|---|
| Initiator | By signing, the author is attesting that the content of the document is complete and accurate. |
| Reviewer | By signing, the reviewer is attesting that the document's approach and contents are compliant with the study protocol, all appropriate, regulatory requirements, and other significant guidelines. This individual(s) has reviewed the document for accuracy and completeness. |

# **TABLE OF CONTENTS**

| 1 | Introduction | 8 |
|---|---|---|
| 2 | Study Objective | 8 |
| 3 | Study Design | 8 |
| 4 | Endpoints | 8 |
| 4.1 | Primary Efficacy Endpoint. | 8 |
| 4.2 | Secondary Efficacy Endpoints | 8 |
| 4.3 | Safety Assessments | 9 |
| 5 | General Statistical Considerations | 9 |
| 5.1 | Statistical Methodology | 9 |
| 5.2 | Analysis Populations | 10 |
| 5.2.1 | Intent-to-Treat (ITT) Population | 10 |
| 5.2.2 | Safety Population. | 10 |
| 5.3 | Data Handling Rules and Presentation Specifications | 10 |
| 6 | Subject Accountability and Disposition. | 11 |
| 7 | Demographics and Baseline Characteristics | 11 |
| 7.1 | Demographics and Important Baseline Characteristics | 11 |
| 7.2 | Medical History | 11 |
| 8 | Treatments and Medications | 11 |
| 8.1 | Prior and Concomitant Medications | 11 |
| 8.2 | Study Drug Exposure | 12 |
| 8.3 | Compliance | 12 |
| 9 | Efficacy Analyses | 12 |
| 9.1 | Primary Efficacy Endpoint - Proportion of Subjects who Never Received Mechanical Ventilation and/or ECMO and Alive at Day 28 | 12 |
| 9.2 | Proportion of Subjects Alive, Discharged, and not on Supplemental Oxygen, Proportion Subjects who Never Received Mechanical Ventilation and/ or ECMO and Alive, and Proportion of Subjects Deceased | |
| 9.3 | Time to Recovery, Time to Mechanical Ventilation/ECMO or All-cause Mortality, and Time to death | 13 |
| 9.4 | Clinical Status Based on the NIAID 8-point Ordinal Scale at Day 28 | 13 |
| 9.5 | Number of Days in ICU/CCU and Number of Days on Mechanical Ventilation and/or ECMO | 14 |

| 9.6 | Change in Categorical PaO <sub>2</sub> /FiO <sub>2</sub> Ratio (Mild, Moderate, and Severe) | 14 |
|---|---|---|
| 9.7 | Change from Baseline in PaO2/FiO2 Ratio and Change from baseline in Resting SpO2/FiO2 at Day 28 | 14 |
| 9.8 | Change in (Non-invasive) Oxygen Supplementation Requirements at Day 28 | 14 |
| 10 | Safety Analyses | 14 |
| 10.1 | Adverse Events | 15 |
| 10.2 | Vital Signs | 15 |
| 10.3 | Laboratory Tests | 15 |
| 11 | Interim Analysis | 15 |
| 12 | Reference | 15 |
| Appe | ndix I Handling Missing/Incomplete Dates | 16 |
| Appe | ndix II Standardized meddra queries (SMQ) for Hypersensitivity reaction | 17 |
| Anne | ndix III Standardized Meddra queries (SMO) for Anaphylactic Reaction | 30 |

#### LIST OF ABBREVIATIONS

**AE** Adverse Event

ALP Alkaline Phosphatase

**ARDS** Acute Respiratory Distress Syndrome

AST Aspartate Aminotransferase

ALT Alanine Aminotransferase

**ANOVA** Analysis of Variance

**AST** Aspartate Aminotransferase

ATC Anatomical Therapeutic Class

BMI Body Mass Index

**BSA** Body Surface Area

CI Confidence Interval

**CRF** Case Report Form

CTCAE Common Terminology Criteria for Adverse Events

CTGF Connective Tissue Growth Factor

DMC Data Monitoring CommitteeDBP Diastolic Blood Pressure

**DMP** Data Management Plan

ECG Electrocardiogram

**EOS** End of Study

**EOT** End of Treatment

**HAHA** Human Anti-Pamrevlumab Antibody

ICH E9 International Conference on Harmonization Statistical Principles for

Clinical Trials

**ITT** Intent-To-Treat

IV Intravenous

LLN Lower Limit of Normal, value provided by the laboratory

MAR Missing At Random

**MedDRA** Medical Dictionary for Regulatory Activities

NIAID National Institute of Allergy and Infectious Diseases

PCS Potentially Clinically Significant

PT Preferred Term

**SMQ** Standardized MedDRA Queries

**SOC** System Organ Class

SAE Serious Adverse Event

**SAP** Statistical Analysis Plan

**SBP** Systolic Blood Pressure

**TEAE** Treatment Emergent Adverse Event

**TESAE** Treatment Emergent Serious Adverse Event

TLF Table, Listing, and Figure

ULN Upper Limit of Normal, value provided by the laboratory

**WHODD** World Health Organization Drug Dictionary

WHO World Health Organization

#### 1 INTRODUCTION

The study was terminated by Sponsor on February 19, 2021. Twenty-two subjects were randomized for the study at the study termination. This statistical analysis plan (SAP) provides a more detailed elaboration of the analyses.

# 2 STUDY OBJECTIVE

To assess the efficacy and safety of intravenous pamrevlumab, an investigational monoclonal antibody against connective-tissue growth factor (CTGF), compared to placebo, in hospitalized patients with acute COVID-19 disease due to confirmed SARS-COV-2 infection.

#### 3 STUDY DESIGN

This is a randomized, double-blind, placebo-controlled phase 2 study of the efficacy and safety of intravenous pamrevlumab, a monoclonal antibody against connective-tissue growth factor (CTGF), in hospitalized subjects with acute COVID-19 disease due to SARS-CoV-2 infection.

Eligible subjects are those with documented SARS-CoV-2 infection, age 40 to 85 years, with evidence of respiratory compromise requiring hospital admission. This age range is chosen to enhance detection of potential clinical benefits in subjects at highest risk for developing severe COVID-19 disease in this proof-of-concept study.

The total sample size is approximately 130 subjects. Subjects are randomized in a 1:1 ratio, according to a pre-determined randomization list from a permuted block design, to receive either pamrevlumab or placebo. All subjects are treated with standard-of-care according to the judgment of the Investigator.

Study drug is administered as IV infusion on Days 1 (day of randomization), 7, 14 and 28. A follow-up visit is performed 4 weeks after the last dose.

#### 4 ENDPOINTS

# 4.1 Primary Efficacy Endpoint

The primary endpoint is the proportion of subjects who never received mechanical ventilation and/or ECMO and alive at Day 28.

# 4.2 Secondary Efficacy Endpoints

- Proportion of subjects alive, discharged home, and not on supplemental oxygen at Day 28
- Proportion of subjects who never received mechanical ventilation and/ or ECMO and alive at Day 14
- Time to recovery by Day 28 based on the NIAID 8-point ordinal scale (Day of recovery is defined as the first day on which the patient satisfies one of the following three

categories from the ordinal scale: (1) Not hospitalized, no limitations on activities; (2)Not hospitalized, limitations on activities and/or requiring home oxygen; (3) Hospitalized, not requiring supplemental oxygen, no longer requiring medical care (used if hospitalization was extended for infection-control reasons)

- Clinical status based on the NIAID 8-point ordinal scale (time range: Days 1 to 28)
- Days in ICU/CCU (either on or off mechanical ventilation and/or ECMO) at Day 28
- Days on mechanical ventilation and/or ECMO at Day 28
- Time to mechanical ventilation/ECMO or all-cause mortality at Day 28
- All-cause mortality at Day 28 (proportion of subjects deceased)
- Time to death from any cause at Day 28
- Change in PaO<sub>2</sub>/FiO<sub>2</sub> ratio as categorical variable using Berlin criteria for ARDS categorization (mild, moderate, severe) (time range: Days 1 to 28)
- Change in PaO<sub>2</sub>/FiO<sub>2</sub> ratio as continuous variable (time range: Days 1 to 28)
- Change in resting SpO<sub>2</sub> adjusted by FiO<sub>2</sub> (time range: Days 1 to 28)
- Change in (non-invasive) oxygen supplementation requirements (time range: Days 1 to 28)

# 4.3 Safety Assessments

Treatment-emergent adverse events (TEAEs); treatment-emergent serious adverse events (TESAEs), including hypersensitivity/ anaphylactic reactions, and vital signs.

#### 5 GENERAL STATISTICAL CONSIDERATIONS

All data collected will be included in the data listings. All analyses will be performed using SAS® Version 9.3 or higher.

#### 5.1 Statistical Methodology

There will be no treatment comparison analysis performed for this early terminated study.

Baseline is defined as the last value on or before the first infusion.

Continuous variables will be summarized using descriptive statistics: n, mean, standard deviation (SD), standard error (SE), median, 25th and 75th percentile, minimum, and maximum. The 2-sided 95% confidence interval for the treatment group mean will be presented as appropriate. Categorical variables will be tabulated by frequency count and percentage. The confidence interval for the proportions for each treatment group will be calculated using the Clopper-Pearson method as appropriate.

The Clopper-Pearson exact 95% CIs for the dichotomous parameters will be from SAS FREQ procedures with option BINOMIAL (EXACT). The 95% CIs for means of normally distributed parameters will be from appropriate SAS procedures such as PROC MEANS.

Analyses will be performed using SAS® Version 9.3 or higher.

# 5.2 Analysis Populations

The study population is defined through inclusion/exclusion criteria to reflect the targeted patient population for study. The details of the inclusion/exclusion criteria can be found in the protocol.

### 5.2.1 Intent-to-Treat (ITT) Population

The ITT population is defined as all randomized subjects. Subjects will be analyzed according to the treatment as randomized.

### **5.2.2** Safety Population

The safety population is defined as all subjects who have received any study medication. Subjects will be analyzed according to the treatment as received.

# 5.3 Data Handling Rules and Presentation Specifications

The following general guidelines will apply to all statistical analyses and data presentations:

- Age (Years) = INTCK('YEAR', Birth Date, Date of Informed Consent,'C') where INTCK is a SAS function. Age groups are 18 to 64, 64 to 75, >=75
- Duration of Ventilation will be calculated as Ventilation Stop Date/Time –
  max(Ventilation Start Date/Time, Randomization Date [we will use 12:00 if no time
  available] or 1st Dose completion Date/Time)
- All reporting values (mean, SD, 95% CI, etc.) for continuous variables will have the same decimal places as the raw data.
- All percentages will be rounded to one decimal place and lined up by the decimal place. The percentage will be suppressed when the count is zero. All analysis statistics will have the same decimal place as the raw value. All duration of time will have 1 decimal place.
- Body weight, height and temperatures will be converted using the following formula:
  - kg = 1b/2.2- cm = 2.54 x in
  - ${}^{\circ}C = (5/9) \times ({}^{\circ}F 32)$
- Computation formulas:

BSA = [Weight 
$$^{0.425}$$
 (kg) \* Height  $^{0.725}$  (cm)] x .007184  
BMI = Weight (kg) / (Height (m))<sup>2</sup>

- Mean Arterial Pressure (MAP) will be derived using the following equation:
   MAP = (2/3) \* DBP + (1/3) SBP
- For continuous variables that are recorded as "<X" or ">X", the value of "X" will be used in the calculation of summary statistics.
- All tables and listings will have a header showing "FibroGen, Inc.", the protocol number, date of the database transfer, and Page x of y. A footer will show the program file path/name, output file path/name, run date and run time.

# **6** SUBJECT ACCOUNTABILITY AND DISPOSITION

The number and percentage of subjects who are randomized, dosed, treatment prematurely discontinued, and completed the study will be summarized by treatment group. Reasons for premature discontinuation as recorded on the Study Disposition page of the CRF will be summarized.

#### 7 DEMOGRAPHICS AND BASELINE CHARACTERISTICS

### 7.1 Demographics and Important Baseline Characteristics

Demographic parameters and important baseline characteristics will be summarized for ITT population by treatment arm. These include but are not be limited to age, age group, sex, ethnicity, race, weight, body-mass index (BMI), smoking status, and selective medical history.

Descriptive statistics (n, mean, standard deviation, median, 25-75<sup>th</sup> percentiles, minimum, and maximum) will be presented for continuous variables. Frequency distributions (number and percentage of subjects) will be presented for categorical variables.

Descriptive statistics of baseline efficacy assessments will be presented in their change from baseline tables.

### 7.2 Medical History

Medical history will be listed for the Safety population.

# 8 TREATMENTS AND MEDICATIONS

#### 8.1 Prior and Concomitant Medications

The use of the prior and concomitant medications will be listed for the ITT population. The version of WHODRUG used to code the medication is stated in the data management plan (DMP).

Medications are classified into 2 categories:

1. Prior medications - medications that are stopped prior to the first study drug infusion

2. Concomitant medications - medications that are used concomitantly with the study drug, which includes all medications that started after or not stopped before the first infusion.

# 8.2 Study Drug Exposure

Duration of study drug exposure in days is calculated as: (last dose date – first dose date + 1). Duration of study drug exposure will be summarized as a continuous variable. The duration will also be tabulated by the following categories for the Safety population.

```
1 to 3 days
>3 to <=7 days
>7 to <=14 days
>14 days <=21 days
>21 days
```

Pamrevlumab infusion dose (in mg and mg/Kg), number of infusions during study, and interruptions during infusion and reason for interruptions will also be listed.

# 8.3 Compliance

The compliance will be presented as % of actual doses of infusion administered over the expected total dose of infusions during study for the safety population. That is, compliance = actual doses received / scheduled doses \* 100%. Treatment compliance will be listed only.

# 9 EFFICACY ANALYSES

Efficacy data will be summarized descriptively based on observed data for the ITT population. There will be no imputation performed for the missing endpoint value.

# 9.1 Primary Efficacy Endpoint - Proportion of Subjects who Never Received Mechanical Ventilation and/or ECMO and Alive at Day 28

Proportion of subjects never received mechanical ventilation and/or ECMO and alive at Day 28 will be summarized based on observed data.

# 9.2 Proportion of Subjects Alive, Discharged, and not on Supplemental Oxygen, Proportion of Subjects who Never Received Mechanical Ventilation and/or ECMO and Alive, and Proportion of Subjects Deceased

Proportion of subjects alive, discharged home, and not on supplemental oxygen at Day 28, proportion of subjects never received mechanical ventilation and/ or ECMO and alive at Day 14, and proportion of all-cause deaths at Day 28 will be summarized descriptively based on observed data.

# 9.3 Time to Recovery, Time to Mechanical Ventilation/ECMO or All-cause Mortality, and Time to death

• Time (number of days) from randomization to recovery by Day 28 based on NIAID 8-point ordinal scale where recovery is defined as the first day on which the patient satisfies one of the following three categories from the ordinal scale: (1) Not hospitalized, no limitations on activities; (2) Not hospitalized, limitations on activities and/or requiring home oxygen; (3) Hospitalized, not requiring supplemental oxygen, no longer requiring medical care (used if hospitalization was extended for infection-control reasons)

Subjects without the event will be censored at the date of last NIAID 8-point ordinal scale assessment.

• Time (number of days) from randomization to mechanical ventilation/ECMO or all-cause mortality by Day 28

For subjects who did not have the event, the last known assessment date of mechanical ventilation/ECMO use or survival status, whichever later will be defined as the censoring date.

• Time (number of days) from randomization to death from any cause by Day 28

For subjects who are alive, the recorded date of last known alive, last contact date, or the date of the last clinic visit, whichever latest will be defined as the censoring date.

The number of days of the above endpoints will be summarized descriptively as appropriate.

#### 9.4 Clinical Status Based on the NIAID 8-point Ordinal Scale at Day 28

Proportion of subjects by response category on the NIAID 8-point ordinal scale will be summarized descriptively based on observed data at baseline and Day 28.

| Order | Ordinal Level |
|-------|------------------------------------------------------------|
| 1 | Not hospitalized, no limitations on activities |
| 2 | Not hospitalized, limitations on activities and/or |
| | requiring home oxygen |
| 3 | Hospitalized, not requiring supplemental oxygen, no |
| | longer requiring medical care (used if hospitalization was |
| | extended for infection-control reasons) |
| 4 | Hospitalized, not requiring supplemental oxygen, |
| | requiring ongoing medical care (COVID-19-related or |
| | otherwise) |
| 5 | Hospitalized, requiring supplemental oxygen |
| 6 | Hospitalized, requiring high-flow oxygen, non-invasive |
| | mechanical ventilation, or both |

| Statistical Analysis Plan, Version 1.0 |
|----------------------------------------|
|----------------------------------------|

| 7 | Hospitalized, requiring invasive mechanical ventilation, |
|---------|----------------------------------------------------------|
| | extra-corporeal membrane oxygenation (ECMO), or both |
| 8 | Death |
| Missing | |

# 9.5 Number of Days in ICU/CCU and Number of Days on Mechanical Ventilation and/or ECMO

Total number of days in ICU/CCU (either on or off mechanical ventilation and/or ECMO) at Day 28 and total number of days on mechanical ventilation and/or ECMO at Day 28 will be summarized descriptively.

# 9.6 Change in Categorical PaO<sub>2</sub>/FiO<sub>2</sub> Ratio (Mild, Moderate, and Severe)

PaO2/FiO2 ratio will be defined as a categorical variable using Berlin criteria for ARDS categorization (mild, moderate, severe), where mild is PaO2/FiO2 from >200 to <=300, moderate is from 100 to <=200, and severe is <100. Proportion of subjects of each category at baseline and Day 28 will be summarized descriptively.

# 9.7 Change from Baseline in PaO2/FiO2 Ratio and Change from baseline in Resting SpO2/FiO2 at Day 28

Change from baseline in PaO2/FiO2 ratio at Day 28 and change from baseline in resting SpO2 adjusted by FiO2 (SpO2/FiO2) at Day 28 will be summarized descriptively.

#### 9.8 Change in (Non-invasive) Oxygen Supplementation Requirements at Day 28

The non-invasive oxygen supplementation requirements include:

- (1) No oxygen supplementation (including breathe room air or have been discharged from hospital)
- (2) Non-invasive oxygen supplementation -nasal cannula and face-mask

Change in non-invasive oxygen supplementation requirements will be presented by proportion of subjects with non-invasive oxygen supplementation requirements at baseline and at Day 28.

#### 10 SAFETY ANALYSES

The safety analyses will be based on the Safety population.

#### **10.1 Adverse Events**

Adverse events will be coded using the latest Medical Dictionary for Regulatory Activities (MedDRA), and the final version will be stated in the data management plan (DMP). Per protocol, the 28 days after the last dose is the last safety follow up. Therefore, the treatment emergent adverse event (TEAE) is defined as an adverse event (AE) with an onset date on or after the first infusion up to within 28 days from the last infusion date. An AE with missing start date/time will be considered to be a TEAE.

The number (%) of subjects reporting TEAEs in each treatment group will be summarized by system organ class and preferred term; by system organ class, preferred term, and severity; and by system organ class, preferred term, and relationship to study medication. If more than one event occurs with the same SOC/preferred term for the same patient, the patient will be counted only once for that SOC/preferred term using the most severe and most related occurrence for the summarization by severity and by relationship to the study medication.

In addition, number (%) of subjects with treatment-emergent serious AEs (TESAE), number (%) of subjects with non-serious TEAE, number (%) of subjects with most frequent (non-serious) TEAE (>=5%), and number (%) of subjects with TEAE leading to discontinuation will be summarized by SOC/preferred term. The hypersensitivity and anaphylactic reactions will be listed.

Listings of subjects with serious adverse events (SAEs), subjects with adverse events leading to discontinuation, and subjects who died will be provided.

#### 10.2 Vital Signs

The pre- and post-infusion vital signs (systolic and diastolic blood pressure (mmHg), respiration rate (breath/min), heart beat (beat/min), Temperature (C) will be listed for the safety population.

#### 10.3 Laboratory Tests

No laboratory test results were collected.

#### 11 INTERIM ANALYSIS

The study do not have interim analysis.

#### 12 REFERENCE

E9 (R1) Statistical Principles for Clinical Trials: Addendum: Estimands and Sensitivity Analysis in Clinical Trials

#### APPENDIX I HANDLING MISSING/INCOMPLETE DATES

A. Handling Missing/Incomplete AE Onset Date

If the AE onset date is incomplete or missing, the following rules will be applied to impute AE onset date.

- If year and month are present, only day is missing,
  - a) If AE onset Year/month = Day 1 Year/month, assign onset day = day of Day 1 (Day 1 is the first infusion day);
  - b) If AE onset Year/month  $\neq$  Day 1 Year/month, assign onset day = 1<sup>st</sup> of the month;
- If year is present, month and day are missing, or when only month is missing (treating day as missing),
  - a) If AE onset year = year of Day 1, assign onset date = month and day part of Day 1 date:
  - b) If AE onset year  $\neq$  year of Day 1, assign onset date= January 1<sup>st</sup>.
- If onset date is completely missing, assign onset date = date of Day 1.

If the stop date is complete and the imputed start date as above is after the stop date, the start date will be imputed by the stop date.

# B. Handling Missing/Incomplete Prior or Concomitant Medication Start/Stop Dates

For prior or concomitant medications, including rescue medications, incomplete (i.e., partially missing) start date is imputed the same way as for the AE described above. When the start date and the stop date are both incomplete for a patient, impute the start date first.

# **Incomplete Stop Date**

The following rules are applied to impute the missing stop date, if needed.

- If year is present, month and day are missing, or when only month is missing (treating day as missing)
  - a) If stop year = year of last dose, assign stop date = month and day of the last dose date;
  - b) If stop year  $\neq$  year of Day 1, assign stop date= December 31<sup>st</sup>.
- If year and month are present, only day is missing,
  - a) If AE stop Year/month = Year/month of last dose date, assign stop day = day part of last dose date
  - b) If AE stop Year/month \neq Day 1 Year/month, assign onset day = last day of the month:
- Impute CM end date even if 'ONGOING' is checked so as to report the CM treatment duration in the study if needed.

# APPENDIX II STANDARDIZED MEDDRA QUERIES (SMQ) FOR HYPERSENSITIVITY REACTION


FG-CLPLN-0010

FGCL-3019-098 Statistical Analysis Plan, Version 1.0 04/20/021

| Wheezing | 10047924 | Broad | 16.0 | 16.0 |
|----------|----------|-------|------|------|

# APPENDIX III STANDARDIZED MEDDRA QUERIES (SMQ) FOR ANAPHYLACTIC REACTION


# Document Approvals Approved Date(GMT-08:00): 03 May 2021

| Approval Task<br>Verdict: Approve | 26-Apr-2021 18:54:34 GMT+0000 |
|-----------------------------------|-------------------------------|
| Approval Task<br>Verdict: Approve | 26-Apr-2021 19:15:40 GMT+0000 |
| Approval Task<br>Verdict: Approve | 26-Apr-2021 19:45:49 GMT+0000 |
| Approval Task<br>Verdict: Approve | 28-Apr-2021 00:32:57 GMT+0000 |
| Approval Task<br>Verdict: Approve | 28-Apr-2021 00:52:26 GMT+0000 |

# Document Approvals Approved Date(GMT-08:00): 03 May 2021

| Approval Task<br>Verdict: Approve | |
|-----------------------------------|-------------------------------|
| | 03-May-2021 15:39:26 GMT+0000 |